CLINICAL TRIAL: NCT04016194
Title: Multiple-breath Washout for Lung Function Testing in Children With Cystic Fibrosis: Predictive for Survival?
Brief Title: Prediction of Survival in Children With Cystic Fibrosis Using the Multiple-breath Washout
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Lindenhofspital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 3840
Record Dates: First submitted 2019-05-07; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Cystic Fibrosis; Death; Lung Transplantation
Keywords: Multiple-breath washout, MBW; Lung clearance index, LCI; Prediction; Survival; Cystic Fibrosis, CF
MeSH Terms: conditions — Cystic Fibrosis; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lung function testing — Multiple-breath washout (MBW) is a safe, easy and sensitive lung function test using inert gases such as Nitrogen (N2) to assess efficiency of ventilation distribution. The latter can be estimated by the lung clearance index (LCI), an established study end-point in patients with CF
  Other Names: Multiple-breath washout, MBW

SUMMARY:
Retrospective cohort study using routinely collected annual data on lung clearance index (LCI) in combination with clinical data to predict survival in patients with Cystic Fibrosis. The primary study endpoint is the association of LCI with the compound outcome survival or lung transplantation in patients with CF.

DETAILED DESCRIPTION:
Retrospective analysis of longitudinal data collected during clinically routine from approximately 200 patients with CF aged 3 years or more between 01.01.1980 and 31.12.2005. The overall aim of this project is to retrospectively assess whether LCI measured for clinical purposes during school age is predictive for survival or lung transplantation in adulthood. For this, the investigators will assess in a systematic way clinically measured LCI and relate them with the compound outcome survival or lung transplantation retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated at the Children's Hospital Bern
* Confirmed CF Diagnosis
* Age >= 3 years

Exclusion Criteria:

* Uncertain diagnosis of CF according to current standards
* Existing written or otherwise documented refusal to participate in research

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-Probability sample
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 1990-01-01 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Lung clearance index (LCI) | Lung function is collected quarterly until outcome (death or lung transplantation) or end of Study (12/2005) is reached
  Lung function outcome derived by MBW and the compound Outcomes mortality or lung transplantation

SECONDARY OUTCOMES:
Functional residual capacity (FRC) | Lung function is collected quarterly until outcome (death or lung transplantation) or end of Study (12/2005) is reached
  Lung function outcome derived by MBW
Forced expired Volume in 1 second (FEV1) | Lung function is collected quarterly until outcome (death or lung transplantation) or end of Study (12/2005) is reached
  Lung function outcome derived by Spirometry
Body weight | Characteristics are collected quarterly until outcome (death or lung transplantation) or end of Study (12/2005) is reached
  Anthropometric characteristics
Body length | Characteristics are collected quarterly until outcome (death or lung transplantation) or end of Study (12/2005) is reached
  Anthropometric characteristics
Gender | Characteristics are collected quarterly until outcome (death or lung transplantation) or end of Study (12/2005) is reached
  Anthropometric characteristics
Presence of Pseudomonas aeruginosa infection | Characteristics are collected quarterly until outcome (death or lung transplantation) or end of Study (12/2005) is reached
  Clinical characteristics
Presence of Staphylococcus aureus infection | Characteristics are collected quarterly until outcome (death or lung transplantation) or end of Study (12/2005) is reached
  Clinical characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Florian Singer, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (2):
- Switzerland (2):
  - University Children's Hospital Bern, Bern
  - Lindenhof Spital, Quartier Bleu, Bern

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with researchers involved in the data collection and analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Until 12/2020
Access Criteria: Researchers involved in data collection

REFERENCES:
- [Derived] Kurz JM, Ramsey KA, Rodriguez R, Spycher B, Fischer Biner R, Latzin P, Singer F. Association of lung clearance index with survival in individuals with cystic fibrosis. Eur Respir J. 2022 Mar 3;59(3):2100432. doi: 10.1183/13993003.00432-2021. Print 2022 Mar. PMID 34289977